CLINICAL TRIAL: NCT03468998
Title: A Randomized Trial to Evaluate the Effect of Allograft Bone Particle Size on Histomorphometric and Clinical Outcomes Following Ridge Preservation/Augmentation Procedures
Brief Title: The Influence of Bone Allograft Particle Sizes on the Quantity and Quality of New Bone Formation in Grafted Extraction Sockets and Edentulous Ridges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Ramzi V. Abou-Arraj, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RAP-17
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Alveolar Ridge Augmentation; Alveolar Ridge Preservation
Keywords: Bone allograft; Particle size; Ridge preservation; Ridge augmentation; Socket grafting; Histology; New bone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Ridge Preservation with Small Particle Allograft (Active Comparator)
  Interventions: Device: Socket Grafting with small particle allograft
- Ridge Preservation with Large Particle Allograft (Active Comparator)
  Interventions: Device: Socket Grafting with large particle allograft
- Ridge Augmentation with Small Particle Allograft (Active Comparator)
  Interventions: Device: Lateral ridge augmentation with small particle allograft
- Ridge Augmentation with Large Particle Allograft (Active Comparator)
  Interventions: Device: Lateral ridge augmentation with large particle allograft

INTERVENTIONS:
Device: Socket Grafting with small particle allograft — Small Particle Bone Allograft of 0.25-1.0 mm placed in extraction socket
  Arms: Ridge Preservation with Small Particle Allograft
Device: Socket Grafting with large particle allograft — Large Particle Bone Allograft of 1.0-2.0 mm placed in extraction socket
  Arms: Ridge Preservation with Large Particle Allograft
Device: Lateral ridge augmentation with small particle allograft — Small Particle Bone Allograft of 0.25-1.0 mm used in lateral ridge augmentation (Guided Bone Regeneration) and covered with a collagen membrane
  Arms: Ridge Augmentation with Small Particle Allograft
Device: Lateral ridge augmentation with large particle allograft — Large Particle Bone Allograft of 1.0-2.0 mm used in lateral ridge augmentation (Guided Bone Regeneration) and covered with a collagen membrane
  Arms: Ridge Augmentation with Large Particle Allograft

SUMMARY:
This study will evaluate the effect of allograft bone particle size on the bone quantity and quality following socket grafting and lateral ridge augmentation in preparation for endosseous implant placement.

Pre (baseline)- and post-grafting (3 months for sockets and 6 months for edentulous ridges) clinical as well as 2- and 3-dimensional radiographic measurements will be used to evaluate the differences between sites grafted with small vs. large particle sized bone allografts.

Histological analysis will be performed at time of surgical re-entry of grafted sites to place the dental implants, and assessed for differences in new bone formation between the 2 types of grafts.

DETAILED DESCRIPTION:
This study is a prospective, two-arm, randomized trial that will evaluate and compare the bone healing following ridge preservation of extraction sockets (RP, Arms 1 and 2) or lateral ridge augmentation of edentulous sites (RA, Arms 3 and 4) using either small particle (SP) or large particle (LP) mineralized cortico-cancellous bone allografts in a total of 48 patients (12 in each arm).

Study approval was obtained from the university's institutional review board. Qualifying participants and defects are randomized following a computerized permutation block to receive either LP or SP allografts on day of surgery. In the RP arms, tooth extraction is performed with a flapless minimally invasive technique, followed by socket grafting with a randomized graft covered with a collagen dressing and sutures. In the RA arms, lateral ridge augmentation is conducted utilizing a randomized bone graft covered by a collagen membrane fixated with tacks.

The mineralized cortico-cancellous bone allografts utilized in this study were all obtained from the same donor, lot and tissue bank to account for variation in age, race, gender and related healing potential of different graft sources.

In the RP arm, bone core biopsies will be harvested at time of implant placement 3 months following socket grafting, whereas similar biopsies will be obtained at 6 months following lateral ridge augmentation in the RA group. These 2x2x6 mm bone cores will then undergo histological and histomorphometrical analyses to determine qualitative and quantitative healing differences between LP and SP in all study arms.

Clinical measurements are gathered at 2 time points (grating and implant placement) at all defects and will be compared for differences.

Cone beam computed tomography (CBCT) initial scans are conducted immediately following socket grafting (RP arms) and prior to ridge augmentation (RA arms) and second scans obtained prior to implant placement (all RP and RA arms). Virtual implant planning software (coDiagnostiX) will be utilized to assess and compare the 2- and 3-dimensional changes for all defects.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 18 years old
* Must be a patient of the UAB Dental School
* Able to read and understand informed consent document
* Need for implants to replace missing tooth or teeth in at least one quadrant of the mouth.
* Hopeless tooth or teeth planned to be replaced with dental implant(s)_socket with residual 4 walls following minimally invasive tooth extraction (a dehiscence of <3mm may be included) or insufficient alveolar ridge width for endosseous implant placement defined as 5mm or less as determined by bone sounding and cone beam computed tomography (CBCT) scan.
* Patient and/or guardian is willing and able to comply with the preoperative and postoperative diagnostic and clinical evaluations required.

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old
* Smokers/tobacco users (>10 cigarettes/day)
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Patients with significant medical conditions or habits expected to interfere with bony healing.
* Patient is a poor compliance risk (i.e., poor oral hygiene, history of alcohol or drug abuse)
* Bone dehiscence of >4mm following tooth extraction or Vertical loss of bone at edentulous ridge

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi V Abou-Arraj, DDS, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomization was performed by site in the mouth to receive either Small Particle (SP) or Large Particle (LP) Allograft. As a result, some participants received only one of the 2 interventions if they only had one qualifying site while other participants received both interventions if they had multiple sites that met the inclusion criteria in either of the study arms.
  Ridge Preservation: # of SP sites=8 & # of LP sites=7. Ridge Augmentation: # of SP sites=7 & # of LP sites=12 .
Units Other Than Participants: Sites
Groups:
- Ridge Preservation With Small & Large Particle Allograft: This arm applies to patients who had more than 1 qualifying site for ridge preservation. Those sites were randomized to either small or large particles.
- Ridge Augmentation With Small & Large Particle Allograft: This arm applies to patients who had more than 1 qualifying site for ridge augmentation. Those sites were randomized to either small or large particles.
Period: Overall Study
Arm/Group | Ridge Preservation With Small Particle Allograft | Ridge Preservation With Large Particle Allograft | Ridge Preservation With Small & Large Particle Allograft | Ridge Augmentation With Small Particle Allograft | Ridge Augmentation With Large Particle Allograft | Ridge Augmentation With Small & Large Particle Allograft
Started | 7; 8 Sites | 7; 7 Sites | 1; 2 Sites | 10; 10 Sites | 10; 10 Sites | 2; 4 Sites
Completed | 6; 7 Sites | 6; 6 Sites | 1; 2 Sites | 6; 6 Sites | 9; 9 Sites | 2; 4 Sites
Not Completed | 1; 1 Sites | 1; 1 Sites | 0; 0 Sites | 4; 4 Sites | 1; 1 Sites | 0; 0 Sites
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Sites
Groups:
- Total: Total of all reporting groups
Arm/Group | Ridge Preservation With Small Particle Allograft | Ridge Preservation With Large Particle Allograft | Ridge Preservation With Small & Large Particle Allograft | Ridge Augmentation With Small Particle Allograft | Ridge Augmentation With Large Particle Allograft | Ridge Augmentation With Small & Large Particle Allograft | Total
Number analyzed (Participants) | 6 | 6 | 1 | 6 | 9 | 2 | 30
Number analyzed (Sites) | 7 | 6 | 2 | 6 | 9 | 4 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 1 | 3 | 4 | 0 | 13
  >=65 years | 5 | 2 | 0 | 3 | 5 | 2 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 1 | 4 | 5 | 1 | 16
  Male | 4 | 3 | 0 | 2 | 4 | 1 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 2
  White | 6 | 6 | 1 | 5 | 8 | 2 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: New Bone Formation (in %) With the Use of Small vs. Large Particle Bone Allografts
Description: Compare histomorphometric amount of new bone formation (in %) between small and large particle bone allografts following ridge preservation and ridge augmentation procedures using core biopsies harvested at time of dental implant placement.
Time Frame: 3 months following socket preservation and 6 months following ridge augmentation
Measure: Mean (Standard Deviation); unit: % of new bone
Units Other Than Participants: Sites
Arm/Group | Ridge Preservation With Small Particle Allograft | Ridge Preservation With Large Particle Allograft | Ridge Augmentation With Small Particle Allograft | Ridge Augmentation With Large Particle Allograft
Number analyzed (Participants) | 7 | 7 | 7 | 11
Number analyzed (Sites) | 8 | 7 | 7 | 12
% of new bone | 17.3 (12.8) | 25.9 (9.5) | 41.0 (10.1) | 31.4 (14.8)

2. Secondary Outcome: Radiographic Ridge Dimensional Changes (in mm) as a Result of Ridge Preservation and Ridge Augmentation Using Small vs. Large Particle Allograft
Description: Using cone beam computed tomography and implant planning software, the bucco-lingual ridge width is measured (in mm) relative to a fixed digital reference and compared between the 2 bone particle groups
Time Frame: from time of grafting until implant placement (3 months following ridge preservation and 6 months following ridge augmentation)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Sites
Arm/Group | Ridge Preservation With Small Particle Allograft | Ridge Preservation With Large Particle Allograft | Ridge Augmentation With Small Particle Allograft | Ridge Augmentation With Large Particle Allograft
Number analyzed (Participants) | 7 | 7 | 7 | 11
Number analyzed (Sites) | 8 | 7 | 7 | 12
mm | 1.1 (0.7) | 0.8 (0.5) | 3.7 (1.3) | 5.1 (1.7)

ADVERSE EVENTS:
Time Frame: From baseline to 3 months following ridge preservation and from baseline to 6 months following ridge augmentation
Arm/Group | Ridge Preservation With Small Particle Allograft | Ridge Preservation With Large Particle Allograft | Ridge Preservation With Small & Large Particle Allograft | Ridge Augmentation With Small Particle Allograft | Ridge Augmentation With Large Particle Allograft | Ridge Augmentation With Small & Large Particle Allograft
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/1 | 0/6 | 0/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/1 | 0/6 | 0/9 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/1 | 0/6 | 0/9 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT03468998/Prot_SAP_001.pdf